CLINICAL TRIAL: NCT05341128
Title: Patient Characteristics, Treatment Patterns, and Resource Usage in Children Diagnosed With Central Precocious Puberty (CPP) in China
Brief Title: A Study of Medical Records From Children With Central Precocious Puberty (CPP) in China
Acronym: PACTURE
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: Leuprorelin-5007
Record Dates: First submitted 2022-04-18; First posted 2022-04-22 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Central Precocious Puberty
Keywords: Central Precocious Puberty
MeSH Terms: conditions — Puberty, Precocious

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All Participants With CPP: Pediatric participants who have been diagnosed with CPP, who are currently or previously undergoing with gonadotropin-releasing hormone agonist (GnRHa) treatment between 2015, and 31 December 2024 will be assessed retrospectively using the Chinese CPP Big Data Platform database.

SUMMARY:
The main purpose is to describe how many children were treated during 24 months or less because of CPP and how treatment worked for them.

There are no participants in this trial, the study only involves reviewing participants medical past and current records and collecting information.

DETAILED DESCRIPTION:
This is an observational, non-interventional, retrospective study to evaluate the participants characteristics, current treatment patterns and resource usage in Chinese pediatric participants diagnosed with CPP.

This study will enroll approximately 1000 participants.

The data available in an existing data source the Chinese CPP Big Data Platform database will be analyzed. All the participants will be assigned to a single observational cohort:

• Pediatric Participants With CPP

This multi-center trial will be conducted in China. The overall duration of the study will be approximately 3 years.

ELIGIBILITY:
Inclusion Criteria:

• Participants diagnosed with CPP and treated with GnRHa from the centers participating in this study within the Chinese CPP Big Data Platform database since 2015 to 2024.

CPP diagnosis is based on the clinical assessment and description by CPP specialized doctors.

Exclusion Criteria:

* Not received GnRHa as the treatment for CPP.
* No available data for analysis.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric participants with a diagnosis of CPP who are currently or previously undergoing GnRHa treatment between 2015 and 31 December 2024 will be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 1477 (Actual)
Dates: Start 2023-12-13 (Actual); Primary Completion 2025-08-27 (Actual); Study Completion 2025-08-27 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With CPP Treatment | Up to approximately 10 years

SECONDARY OUTCOMES:
Percentage of Participants With CPP Treatment at Baseline | At Baseline
Percentage of Participants With Luteinizing hormone (LH) Suppression | Baseline up to approximately 10 years
Percentage of Participants With Treatment-emergent Adverse Events (TEAEs) | Up to approximately 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (5):
- China (5):
  - The Second Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Hainan Women and Children's Medical Center, Haikou, Hainan
  - Tongji Hospital affiliated to Tongji Medical College of Huazhong University of Science & Technology, Wuhan, Hubei
  - Shandong Provincial Hospital Affiliated to Shandong First Medical University, Jinan, Shandong
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: Click here for more information about this trial in easy-to-understand language. — https://clinicaltrials.takeda.com/study-detail/88f831d40d9d43b3??page=1&idFilter=Leuprorelin-5007